CLINICAL TRIAL: NCT02553343
Title: Safety and Immunogenicity Trial of High-Dose Quadrivalent Influenza Vaccine Administered by Intramuscular Route in Subjects Aged 65 Years and Older
Brief Title: A Study of the Safety and Immunogenicity of High-Dose Quadrivalent Influenza Vaccine in Subjects Aged 65 Years and Older
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: QHD01; U1111-1161-2450 (Other: WHO)
Record Dates: First submitted 2015-09-15; First posted 2015-09-17 (Estimated); Last update posted 2018-02-09 (Actual); Status verified 2018-02

CONDITIONS: Influenza
Keywords: Influenza; High-Dose Quadrivalent Influenza Vaccine; High-Dose Trivalent Influenza Vaccine
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- QIV HD1 Group (Experimental): Adults ≥ 65 years of age randomly assigned to receive an intramuscular injection of one dose of High-Dose quadrivalent influenza vaccine (formulation 1)
  Interventions: Biological: High-dose quadrivalent influenza virus vaccine
- QIV HD2 Group (Experimental): Adults ≥ 65 years of age randomly assigned to receive an intramuscular injection of one dose of High-Dose quadrivalent influenza vaccine (formulation 2)
  Interventions: Biological: High-dose influenza virus vaccine
- TIV HD1 Group (Active Comparator): Adults ≥ 65 years of age randomly assigned to receive an intramuscular injection of one dose of licensed High Dose trivalent influenza vaccine
  Interventions: Biological: High-dose trivalent inactivated influenza vaccine
- TIV HD2 Group (Active Comparator): Adults ≥ 65 years of age randomly assigned to receive an intramuscular injection of one dose of investigational High-Dose trivalent influenza vaccine
  Interventions: Biological: High-dose trivalent inactivated influenza vaccine

INTERVENTIONS:
Biological: High-dose quadrivalent influenza virus vaccine — 0.5 mL, Intramuscular (IM), injected into the deltoid area
  Other Names: High-dose quadrivalent influenza virus vaccine (QIV HD1)
  Arms: QIV HD1 Group
Biological: High-dose influenza virus vaccine — 0.5 mL, Intramuscular (IM), injected into the deltoid area
  Other Names: High-dose quadrivalent influenza virus vaccine (QIV HD2)
  Arms: QIV HD2 Group
Biological: High-dose trivalent inactivated influenza vaccine — 0.5 mL, Intramuscular (IM), injected into the deltoid area
  Other Names: Fluzone® High-Dose, TIV HD1
  Arms: TIV HD1 Group
Biological: High-dose trivalent inactivated influenza vaccine — 0.5 mL, Intramuscular (IM), injected into the deltoid area
  Other Names: TIV HD2
  Arms: TIV HD2 Group

SUMMARY:
The aim of the study is to assess the safety and immunogenicity of two formulations of the high-dose quadrivalent influenza vaccine compared to the licensed high-dose trivalent influenza vaccine control in healthy elderly subjects aged 65 years of age and above.

Primary objectives:

* To describe the safety profile of all subjects in each study group.
* To demonstrate that the high-dose quadrivalent influenza vaccine induces an immune response (as assessed by HAI geometric mean titers (GMTs) that is non-inferior to responses induced by the licensed high-dose trivalent influenza vaccine for the 3 common virus strains at 28 days post-vaccination.

Secondary objectives:

* To describe post-vaccination immunogenicity for the 4 virus strains (as assessed by seroconversion and seroprotection) for subjects who receive the high-dose quadrivalent influenza vaccine and the licensed high-dose trivalent influenza vaccine.
* To describe post-vaccination immunogenicity for the 4 virus strains (as assessed by GMTs, seroconversion, and seroprotection) for subjects who receive the high-dose quadrivalent influenza vaccine and the investigational high-dose trivalent influenza vaccine.

DETAILED DESCRIPTION:
All eligible participants will be randomized to receive a single injection of either one of the high-dose quadrivalent influenza vaccine formulations or one of the high-dose trivalent influenza vaccines at Day 0. They will provide blood samples for hemagglutination inhibition (HAI) testing. Safety information as solicited, unsolicited reactions, serious adverse events, including adverse events of special interest will be collected in the trial.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 65 years on the day of inclusion
* Informed consent form has been signed and dated
* Able to attend all scheduled visits and to comply with all trial procedures.

Exclusion Criteria:

* Participation at the time of trial enrollment (or in the 4 weeks preceding the trial vaccination) or planned participation during the present trial period in another clinical trial investigating a vaccine, drug, medical device, or medical procedure
* Receipt of any vaccine in the 4 weeks (28 days) preceding the trial vaccination or planned receipt of any vaccine prior to Visit 2
* Vaccination against influenza in the past 6 months
* Receipt of immune globulins, blood or blood-derived products in the past 3 months
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccine used in the trial or to a vaccine containing any of the same substances
* Thrombocytopenia or bleeding disorder, contraindicating IM vaccination based on investigator's judgment
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily
* Substance abuse that, in the opinion of the investigator, might interfere with the trial conduct or completion
* Chronic illness that, in the opinion of the investigator, is at a stage where it might interfere with trial conduct or completion
* Identified as an Investigator or employee of the Investigator or trial center with direct involvement in the proposed trial, or identified as an immediate family member (i.e., parent, spouse) of the Investigator or employee with direct involvement in the proposed trial
* Personal or family history of Guillain-Barré syndrome
* Neoplastic disease or any hematologic malignancy (except localized skin or prostate cancer that is stable at the time of vaccination in the absence of therapy and subjects who have a history of neoplastic disease and have been disease free for ≥ 5 years)
* Known allergy to iodinated radiocontrast media
* Moderate or severe acute illness/infection (according to investigator judgment) on the day of vaccination or febrile illness (temperature ≥ 38.0°C [≥ 100.4°F]). A prospective subject should not be included in the trial until the condition has resolved or the febrile event has subsided.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 792 (Actual)
Dates: Start 2015-09; Primary Completion 2016-04-04 (Actual); Study Completion 2016-04-04 (Actual)

PRIMARY OUTCOMES:
Number of participants reporting solicited injection site and systemic events, unsolicited adverse events and serious adverse events following vaccination with a dose of Fluzone influenza vaccines | Day 0 up to 6 months post-vaccination
  Solicited injection site: Pain, Redness, Swelling, Induration, and Ecchymosis. Solicited systemic reaction: Fever (Temperature), Headache, Malaise, Myalgia, and Shivering. Unsolicited adverse events, including serious adverse events, will also be collected
Hemagglutination inhibition (HAI) antibody titers to influenza virus antigens following vaccination with Fluzone High Dose quadrivalent influenza vaccine or High Dose trivalent influenza vaccine | Day 28 post-vaccination

SECONDARY OUTCOMES:
Seroconversion with respect to vaccine antigens following vaccination with Fluzone High-dose quadrivalent influenza vaccine or High-dose trivalent influenza vaccine | Day 28 post-vaccination
  Seroconversion is defined as either a pre-vaccination titer < 10 (1/dil) and a post-vaccination titer ≥ 40 (1/dil), or a pre-vaccination titer ≥ 10 (1/dil) and a ≥ 4-fold increase in post-vaccination titer at 28 days after vaccination.
Seroprotection with respect to vaccine antigens following vaccination with Fluzone High-dose quadrivalent influenza vaccine or High-dose trivalent influenza vaccine | Day 28 post-vaccination
  Seroprotection is defined as a titer ≥ 40 (l/dil) at pre-vaccination and at 28 days after vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (9):
- United States (9):
  - Milford, Connecticut
  - Coral Gables, Florida
  - Wichita, Kansas
  - St Louis, Missouri
  - Rochester, New York
  - Warwick, Rhode Island
  - Nashville, Tennessee
  - Salt Lake City, Utah
  - West Jordan, Utah

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com